CLINICAL TRIAL: NCT04970732
Title: A Randomized Controlled Study to Evaluate the Effectiveness of Chewing Gum in Improving Abdominal Distension After Lumbar Spine Surgery
Brief Title: Effect of Chewing Gum on Abdominal Distension in Patients After Lumbar Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M2018051
Record Dates: First submitted 2021-07-01; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Lumbar Spondylosis
Keywords: Lumbar degenerate diseases; Postoperative management; Abdominal distension
MeSH Terms: conditions — Spondylosis | interventions — Chewing Gum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The patients in the experimental group returned to the ward for general anesthesia, started to wake up for 2 hours, chewed xylitol gum, and the professional nurses distributed it on time every 2 hours on the operation day, then 3 times / day, 15-20 minutes / time, 2 tablets / time. Body position: lateral position. The first anal exhaust stop chewing, normal sleep at night (8 p.m.), do not chew gum. Gum waste must be identified
  Interventions: Procedure: Gum chewing
- Control group (No Intervention): The control group received routine nursing after surgery.

INTERVENTIONS:
Procedure: Gum chewing — The patients in the experimental group returned to the ward for general anesthesia, started to wake up for 2 hours, chewed xylitol gum, and the professional nurses distributed it on time every 2 hours on the operation day, then 3 times / day, 15-20 minutes / time, 2 tablets / time. Body position: lateral position. The first anal exhaust stop chewing, normal sleep at night (8 p.m.), do not chew gum. Gum waste must be identified
  Arms: Experimental group

SUMMARY:
According to chewing gum can promote the recovery of gastrointestinal function, it is used as an intervention measure for patients after lumbar surgery to evaluate the effect of chewing gum on improving abdominal distension of patients after lumbar surgery, so as to provide basis for the application and promotion of chewing gum in lumbar postoperative nursing

DETAILED DESCRIPTION:
In this study, the patients after lumbar surgery were given chewing gum after anesthesia. The exhaust time, defecation time and the incidence of abdominal distension of the two groups were compared, and the significance of chewing gum in improving abdominal distension after lumbar surgery was discussed

ELIGIBILITY:
Inclusion Criteria:

* The subjects aged 18 years or above were able to chew together;
* Good at listening, speaking, reading and writing;
* Lumbar degenerative disease was definitely diagnosed;
* General anesthesia was used;
* Methods: posterior lumbar decompression, bone graft fusion and internal fixation;
* No history of gum allergy;

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Physical examination | After surgery to discharge, an average of 4 days
  Number of bowel sounds
Time points | After surgery to discharge, an average of 4 days
  First anal exhaust time, first defecation time
Medication | After surgery to discharge, an average of 4 days
  Whether the medication for exhaust and defecation is used. If used, what kind of medicine and the dosage of the medicine.
Incidence of abdominal distension | After surgery to discharge, an average of 4 days
  Incidence of abdominal distension

SECONDARY OUTCOMES:
Oral comfort | After surgery to discharge, an average of 4 days
  Whether the oral comfort is applied.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No